CLINICAL TRIAL: NCT04765228
Title: A Prospective One-arm Study of Pegylated Liposomal Doxorubicin Combined With Anlotinib for Neoadjuvant Treatment of Locally Advanced Soft Tissue Sarcoma
Brief Title: Pegylated Liposomal Doxorubicin Combined With Anlotinib for Neoadjuvant Treatment of Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Chen (Other)
Responsible Party: Sponsor-Investigator, Yong Chen, Chief Physician, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB1912212-12
Record Dates: First submitted 2021-01-08; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Stage III Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — liposomal doxorubicin; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pegylated liposomal doxorubicin + Anlotinib (Experimental): Pegylated liposomal doxorubicin 50mg/m2 intravenous infusion on the first day + Anlotinib 12mg/d orally, medication on days 8-21, one cycle every 21 days, 2~4 cycles
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Anlotinib

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — Pegylated liposomal doxorubicin 50mg/m2 intravenous infusion on the first day + Anlotinib 12mg/d orally, medication on days 8-21, one cycle every 21 days, 2~4 cycles
Drug: Anlotinib — Anlotinib

SUMMARY:
A prospective one-arm study of pegylated liposomal doxorubicin combined with anlotinib for neoadjuvant treatment of locally advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
Tumor angiogenesis is very important in the occurrence and development of soft tissue sarcoma. The current clinical studies of molecularly targeted drugs are focused on the advanced treatment stage of soft tissue sarcoma. Anti-angiogenic drugs are not yet available in the neoadjuvant treatment stage of soft tissue sarcoma. Strong evidence. Therefore, this study aimed to evaluate the safety and effectiveness of pegylated doxorubicin liposomes combined with the anti-angiogenic drug Anlotinib for neoadjuvant treatment of patients with soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with soft tissue sarcoma confirmed by histopathology;
2. Patients with soft tissue sarcoma judged to be stage IIB/III according to the AJCC staging of soft tissue sarcoma, or tumors that are closely related to important blood vessels and important nerves suggested by imaging data;
3. No distant transfer
4. According to the preliminary judgment of the research, patients who can improve the effect of surgery by neoadjuvant treatment;
5. Male or female, aged ≥14 years old and ≤75 years old;
6. ECOG score ≤ 2;
7. The expected survival period is ≥3 months;
8. Adequate hematopoietic function: absolute neutrophil count (ANC) ≥ 1.5×109/L and platelet count ≥ 80×109/L and hemoglobin ≥ 9 g/dL;
9. Sufficient liver function: total bilirubin ≤ upper limit of normal (ULN); AST and ALT ≤ 1.5 times the upper limit of normal (ULN); alkaline phosphatase ≤ 5 times the upper limit of normal (ULN);
10. Adequate renal function: serum creatinine ≤ upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min;
11. Visceral function: LVEF≥50%, the New York Society of Visceral Disease Association (NYHA) has a functional classification of I and II, and there is no unhealed wound on the body;
12. Sign the informed consent form.
13. Women should agree to use contraceptive measures (such as intrauterine device (IUD), contraceptives or condoms) during the study period and within 6 months after the end of the study; serum or urine pregnancy within 7 days before study entry The test is negative and must be a non-lactating patient; men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.
14. The patient voluntarily joined the study, signed an informed consent form, had good compliance, and was able to be followed up by the trial staff.

Exclusion Criteria:

1. Ewing's sarcoma, embryonic rhabdomyosarcoma, acinar rhabdomyosarcoma
2. Pregnant or breastfeeding women, or women who are fertile but have not taken contraceptive measures
3. Existing severe acute infection that has not been controlled; or having purulent or chronic infection, and the wound is protracted
4. Active hepatitis B or C
5. Have a history of other tumors within 5 years before treatment, except for cured cervical carcinoma in situ or skin basal cell carcinoma
6. Those who have participated in other drug clinical trials within 4 weeks
7. Patients with pre-existing severe heart disease, including: congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina, myocardial infarction, severe heart valve disease and refractory hypertension, ventricular tachycardia, ventricular, Patients with atrial fibrillation, second-degree type II or third-degree atrioventricular block, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease requiring medication
8. People with uncontrollable neurological or mental diseases or mental disorders, poor compliance, unable to cooperate and describe the treatment response; primary brain tumors or central nerve metastases have not been controlled, and have obvious intracranial hypertension or neuropsychiatry Symptoms
9. Past severe chronic skin diseases
10. People with bleeding tendency, evidence of hereditary bleeding constitution or coagulopathy
11. Have a clear history of allergy to chemotherapy drugs

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of Cycle 3 (each cycle is 21 days)
  Objective Response Rate

SECONDARY OUTCOMES:
pCR rate | One year after the first intravenous drip
  Pathological complete response rate
PFS | 6 weeks after the first intravenous drip
  Progression free survival
OS | After the first intravenous drip,an average of 3 year through study completion
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China